CLINICAL TRIAL: NCT06705140
Title: A Parallel Group, Phase III, Randomized, Observer Blind, Placebo Controlled, Multi Center, Multinational, Multi Arm Study to Demonstrate Non-inferiority of the Immune Response of a Low Dose Compared to the Standard Dose and to Evaluate the Safety of a Respiratory Syncytial Virus Vaccine in Infants and Toddlers (OPAL)
Brief Title: A Study on the Immunogenicity and Safety of 3 Different Dose Concentrations of a Respiratory Syncytial Virus Vaccine in Infants and Toddlers
Acronym: OPAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAD00015; 2023-509536-26 (Registry Identifier: CTIS); U1111-1298-7338 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: RSV Immunisation
Keywords: RSV; RSVt (RSV toddler and Infant) Vaccine
MeSH Terms: interventions — YM 534

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * Blinding for vaccine group assignment: participants, parents or legally acceptable representatives (LARs), outcome assessors, investigators, laboratory personnel, Sponsor study staff
  * No blinding for study staff who prepare and administer the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: Group 1- (SD RSVt vaccine) (Experimental): Participants will receive 2 intranasal administrations of SD RSVt vaccine
  Interventions: Biological: Standard Dose (SD) RSVt vaccine
- Cohort 1: Group 2-Control (Placebo Comparator): Participants will receive 2 intranasal administrations of placebo
  Interventions: Biological: Placebo
- Cohort 1: Group 3- (HD RSVt vaccine) (Experimental): Participants will receive 2 intranasal administrations of HD RSVt vaccine
  Interventions: Biological: High Dose (HD) RSVt vaccine
- Cohort 1: Group 4-Control (Placebo Comparator): Participants will receive 2 intranasal administrations of placebo
  Interventions: Biological: Placebo
- Cohort 2: Group 1- (LD RSVt vaccine) (Experimental): Participants will receive 2 intranasal administrations of LD RSVt vaccine
  Interventions: Biological: Low Dose (LD) RSVt vaccine
- Cohort 2: Group 2- (SD RSVt vaccine) (Experimental): Participants will receive 2 intranasal administrations of SD RSVt vaccine
  Interventions: Biological: Standard Dose (SD) RSVt vaccine
- Cohort 2: Group 3- (HD RSVt vaccine (Experimental): Participants will receive 2 intranasal administrations of HD RSVt vaccine
  Interventions: Biological: High Dose (HD) RSVt vaccine
- Cohort 2: Group 4-Control (Placebo Comparator): Participants will receive 2 intranasal administrations of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low Dose (LD) RSVt vaccine — Pharmaceutical form:
  Liquid for nasal spray
  Route of administration: Intranasal
  Other Names: 534
  Arms: Cohort 2: Group 1- (LD RSVt vaccine)
Biological: Standard Dose (SD) RSVt vaccine — Pharmaceutical form:Liquid for nasal spray-Route of administration:Intranasal
  Other Names: 534
  Arms: Cohort 1: Group 1- (SD RSVt vaccine); Cohort 2: Group 2- (SD RSVt vaccine)
Biological: High Dose (HD) RSVt vaccine — Pharmaceutical form:Liquid for nasal spray-Route of administration:Intranasal
  Other Names: 534
  Arms: Cohort 1: Group 3- (HD RSVt vaccine); Cohort 2: Group 3- (HD RSVt vaccine
Biological: Placebo — Pharmaceutical form:Liquid for nasal spray-Route of administration:Intranasal
  Arms: Cohort 1: Group 2-Control; Cohort 1: Group 4-Control; Cohort 2: Group 4-Control

SUMMARY:
This study is a Phase III, parallel group, randomized, observer blind, placebo controlled, multi-national, multi-center, multi-arm study to be conducted in 947 healthy children enrolled at 6 months to <22 months of age. The purpose of the study is to evaluate the non-inferiority of the immune response of the lower dose (LD) when compared to the standard dose (SD) respiratory syncytial virus infant and toddler (RSVt) vaccine and the safety of the LD, SD and high dose (HD) vaccine in preterm born children and of the HD vaccine in full term born children administered by intranasal route and compared to placebo.

DETAILED DESCRIPTION:
The study duration is approximately 8 months for each participant, including the 6 months safety follow-up phone call after the second study intervention administration.

ELIGIBILITY:
Inclusion Criteria: -Aged 6 months to < 22 months on the day of inclusion (means from the day of the 6-month birthday to the day before the 22-month birthday. The second vaccine administration should be administered before the study participant has turned 24 months of age).

* Participants who are healthy as determined by medical evaluation including medical history.
* For Cohort 1 and Cohort 2 (contingent upon satisfactory safety profile of the RSVt vaccine in Cohort 1):
* Participant born 28 through 36 weeks of gestation and medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study intervention.
* For Cohort 2:
* Participant born at full term of pregnancy (≥ 37 weeks of gestation). Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances.

Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion.

* History of medically diagnosed wheezing. Children with a history of recurrent wheezing will be excluded. Children with a previous single episode of wheezing may be included if that episode of wheezing was not associated with hospitalization or if does not have a family history of wheezing.
* Any acute febrile illness in the past 48 hours that according to investigator judgment is significant enough to interfere with successful inoculation on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Probable or confirmed ongoing case of viral respiratory infection (including COVID-19, influenza, rhinovirus, etc.) at the time of enrollment. A prospective participant should not be included in the study until the respiratory infection has resolved.
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is HIV infected
  * a person who has received chemotherapy within the 12 months prior to study enrollment
  * a person who has received (within the past 6 months) or is receiving (at the time of enrollment) immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Potential close contact with other immunocompromised individual within 30 days after each vaccination as per investigator's discretion.
* Participant's biological mother's previous receipt or planned administration of an investigational RSV vaccine during pregnancy and/or breastfeeding.
* Receipt or planned receipt of any of the following vaccines prior to enrollment or after the first study intervention administration:

  * Any other intranasal live attenuated vaccine within the 28 days prior to and after Dose 1 study administration
  * Unless given on the day of the first study intervention administration, any other injectable live attenuated vaccines within the 28 days prior to and after. Concomitant receipt on the day of the first study intervention administration is allowed
* Planned receipt of any monoclonal antibody for RSV (such as Nirsevimab or Palivizumab) for the duration of the study.
* Previous receipt of an investigational RSV vaccine or receiving any anti-RSV product (such as ribavirin or RSV immune globulin) at the time of enrollment. Previous receipt of an RSV monoclonal antibody within 6 months prior to the first study vaccine administration.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of intranasal and intra-ocular medications within 3 days prior to study enrollment
* Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 6 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 947 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
RSV A serum neutralizing antibody titers at 28 days post dose 2 (D85) | Day 85
  Antibody titers are expressed as GMT at Day 85
RSV B serum neutralizing antibody titers at 28 days post dose 2 (D85) | Day 85
  Antibody titers are expressed as GMT at Day 85
Presence of unsolicited systemic adverse events (AEs) reported in the 30 minutes after each vaccination | Within 30 minutes after each vaccination
  Number of participants experiencing immediate unsolicited systemic AEs
Presence of solicited administration site reactions within 21 days after each vaccination | Within 21 days after each vaccination
  Number of participants experiencing solicited site reactions
Presence of solicited systemic reactions within 21 days after each vaccination | Within 21 days after each vaccination
  Number of participants experiencing solicited systemic reactions
Presence of unsolicited AEs within 28 days after each vaccination | Within 28 days after each vaccination
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events MAAEs throughout the study | Throughout the study (approximately 8 months)
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) throughout the study | Throughout the study (approximately 8 months)
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) throughout the study | Throughout the study (approximately 8 months)
  Number of participants experiencing AESIs

SECONDARY OUTCOMES:
RSV A serum neutralizing antibody titers at baseline (D01) and D85 | At baseline through Day 85
  Antibody titers are expressed as GMTs at baseline and Day 85
RSV B serum neutralizing antibody titers at baseline (D01) and D85 | At baseline through Day 85
  Antibody titers are expressed as GMTs at baseline and Day 85
RSV serum anti-F Immunoglobulin A (IgA) at baseline (Day01) and D85 | At baseline through Day 85
  Antibody titers are expressed as GMTs at baseline and Day 85
RSV serum anti-F Immunoglobulin G (IgG) at baseline (Day01) and D85 | At baseline through Day 85
  Antibody titers are expressed as GMTs at baseline and Day 85
Presence of RSVt vaccine virus viral shedding in D08 and D64 nasal samples | Day 08 through Day 64
  Measured by quantitative real-time polymerase chain reaction (qRT PCR)
Titer of vaccine virus shedding in D08 and D64 nasal samples | Day 08 through day 64
  Quantified by qRT-PCR

CONTACTS AND LOCATIONS:
Locations (4):
- Investigational Site Number : 2140002, Santo Domingo, Dominican Republic
- Honduras (3):
  - Investigational Site Number : 3400002, San Pedro Sula
  - Investigational Site Number : 3400001, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VAD00015 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26337&tenant=MT_SNY_9011